CLINICAL TRIAL: NCT06745063
Title: Arterial Destiffening Effects of SGLT2 Inhibition in Veterans With Obesity
Acronym: EMPA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CARB-015-24S; 2107866 (Other: Local IRB)
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Vascular Health
MeSH Terms: conditions — Obesity | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: placebo-controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Empagliflozin (Experimental): 12 week treatment with 10mg empagliflozin daily
  Interventions: Drug: Empagliflozin
- Placebo (Placebo Comparator): 12 week treatment with 10mg placebo daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin — 12 week treatment with 10mg empagliflozin daily
  Arms: Empagliflozin
Drug: Placebo — 12 week treatment with 10mg placebo daily
  Arms: Placebo

SUMMARY:
The study will assign participants to take either the medication, empagliflozin or a placebo for 12 weeks. The goal of the study is to determine the effects of empagliflozin on arterial health in Veterans with obesity.

DETAILED DESCRIPTION:
The investigators will employ a double-blinded randomized placebo-controlled trial to determine the effects of 12 weeks of SGLT2 inhibition with empagliflozin (10mg daily), or matching placebo, on arterial stiffness in Veterans with obesity. Fifty Veterans with obesity (BMI 30-45kg/m2), 30-60 years of age, will be recruited from the Harry S. Truman Memorial VA Hospital in Columbia, Missouri.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 30-45 kg/m2
* 30-60 years of age at randomization
* Evidence of arterial stiffening (defined as Carotid femoral PWV>age-predicted) at screening visit (PMID: 20530030)

Exclusion Criteria:

* Unable to provide consent
* Diabetes mellitus
* Uncontrolled hypertension (>180/90mmHg) or systolic <100mmHg at screening visit
* Known history of cardiovascular disease: heart failure, ischemic heart disease, peripheral artery disease or stroke
* Diagnosis of chronic kidney disease
* Active cancer (excluding basal cell carcinoma or stage 1 squamous cell carcinoma of the skin)
* Excessive alcohol consumption (>14 drinks/week for men, >7 drinks/week for women)
* Use of GLP-1 analogs or SGLT2 inhibitors
* Use of hormone replacement therapy
* Use of pharmacological therapy for weight loss
* Body weight changes >10% within the past 6 months
* History of hypersensitivity to nitrates
* History of ketoacidosis
* History of recurrent UTIs or mycotic genital infections
* Use of anticoagulants
* Change in anti-hypertensive medication regimen (if in use) during the last 90 days
* Pregnancy

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Carotid-femoral Pulse Wave Velocity (cfPWV) | baseline (t0), week 4, week 8, week 12
  cfPWV is the gold standard non-invasive index of arterial stiffness. Transit time between carotid and femoral pressure waves is calculated using the foot-to-foot method. cfPWV is calculated as distance traveled by the pulse wave (i.e., femoral location-sternal notch minus sternal notch-carotid location) divided by pulse transit time. All the measurements will be done by the same blinded technician. The goal is to assess changes from baseline when compared to weeks 4,8, and 12 time points.

CONTACTS AND LOCATIONS:
Overall Officials: Jaume Padilla Parellada, PhD, Principal Investigator — Harry S. Truman Memorial, Columbia, MO
Locations (1):
- Harry S. Truman Memorial, Columbia, MO, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No